CLINICAL TRIAL: NCT03016065
Title: Efficacy of Pea Hull Fiber Supplementation on Gastrointestinal Transit in Overweight Children.
Brief Title: Efficacy of Pea Hull Fiber - Phase 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Saskatchewan Pulse Growers (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IRB201602266
Record Dates: First submitted 2017-01-06; First posted 2017-01-10 (Estimated); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pea Fiber (Experimental): Snacks fortified with 10 g of pea hull fiber will be administered for two weeks, followed by a two-week washout, and a two-week period with control snacks.
  Interventions: Dietary Supplement: Pea Fiber
- Control (Placebo Comparator): Control snacks will provided for 2 weeks, followed by a two-week washout, and snacks with 10 g/d of pea fiber for 2 weeks.
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Pea Fiber — Baked goods (2 snacks) with fiber-fortified with 5 g/snack of ground pea hulls
  Arms: Pea Fiber
Dietary Supplement: Control — Baked goods (2 snacks) without added fiber
  Arms: Control

SUMMARY:
The purpose of this randomized, cross-over study is to explore the effects of pea hull fiber on bowel movement frequency, transit time, appetite, gastrointestinal symptoms, microbiota composition and activity.

DETAILED DESCRIPTION:
An 8-week randomized, cross-over study will be carried out to assess the efficacy of pea hull fiber. Participants will complete a 2-week baseline period during which appetite, stool frequency, and stool consistency (transit time) will be collected by an online questionnaire, and participants will collect a single stool. Dietary data (Automated Self-Administered 24-Hour diet recall) will be obtained at baseline and at each study visit. Participants will be randomized on or about day 15 and consume snacks without pea hull fiber for a 2-week control period, and snacks with added pea hull fiber for a 2-week treatment period separated by a 2-week washout period. In both intervention periods, participants will complete daily questionnaires to assess stool frequency and consistency (transit time). An online questionnaire assessing appetite will be administered once per week. The GSRS will be competed at each study visit. During washout periods, the same data will be collected as will be done during the baseline and intervention periods. Participants will be asked to collect one stool during baseline and during weeks 4, 6, and 8 for a total of 4 stools. Stool samples will be analyzed for changes in the microbiota.

ELIGIBILITY:
Inclusion criteria:

* Are willing to have height and weight measured and provide demographic information (e.g. age, race, sex).
* Children age between 8-15 years old.
* Are occasionally constipated.
* Are willing to consume pea hull fiber and control snacks daily each for a 2-week period
* Are willing to complete a daily questionnaire throughout the entire 8-week study.
* Are willing to complete the appetite questionnaire two times per week.
* Are willing to complete the Gastrointestinal Symptom Rating Scale (GSRS) bi-weekly.
* Are willing to be interviewed for Automated Self-Administered 24-Hour-Kids-2014 (ASA24-Kids-2014) one time per 2-week period throughout the study.
* Are willing and be able to provide a valid social security for study payment purposes.

Exclusion criteria:

* Have any known food allergies.
* Are currently taking medications for diarrhea.
* Have taken antibiotics within the past four weeks prior to randomization.
* Have ≥ 6 bowel movements per week
* Are currently taking probiotics supplements and do not want to discontinue a minimum of two weeks prior to the study.
* Have previously or are currently being treated for any gastrointestinal diseases such as (gastric ulcers, Crohn's, Celiac, ulcerative colitis, etc.).

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Change in Modified Bristol Stool Form score | Change from baseline at weeks 4, 6 and 8
  Stool consistency rating by Modified Bristol Stool Form for children

SECONDARY OUTCOMES:
Change in number of bowel movements per week | Change from baseline at weeks 4, 6 and 8
  Stool frequency per week

CONTACTS AND LOCATIONS:
Overall Officials: Wendy J Dahl, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Food Science and Human Nutrition Dept, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No